CLINICAL TRIAL: NCT00855205
Title: Rituximab as a Novel Therapy in Refractory Sarcoidosis: A Prospective Open-
Brief Title: Rituximab for Pulmonary Sarcoidosis
Acronym: RIPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor of Medicine, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14889A; NCT00552318 (obsolete NCT alias)
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Sarcoidosis
Keywords: pulmonary sarcoidosis
MeSH Terms: conditions — Sarcoidosis; Sarcoidosis, Pulmonary | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment with rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab will be administered by IV infusion at a dose of 1000 mg (1 g) on day 1 and 15

SUMMARY:
Sarcoidosis is a inflammatory disease affecting many parts of the body, especially the lungs. While most patients do well, there is a group of patients who require continuous doses of prednisone or other drugs. The current study will determine the role of Rituximab as new agent for patients with refractory disease.

DETAILED DESCRIPTION:
Patients with refractory pulmonary sarcoidosis will be eligible for participation in this open label trial of Rituximab as additional therapy. The study will evaluate the efficacy of rituximab in improving the symptoms and functional capacity in patients with chronic sarcoidosis with pulmonary involvement who are symptomatic despite current treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women > 18 years of age.
2. Sarcoidosis diagnosed at least 1 year prior to screening.
3. Histological proven sarcoidosis prior to screening.
4. Have a diagnosis of severe sarcoidosis with evidence of parenchymal disease on chest radiograph (Stage III) or abnormal PFT, with histologic and there should be an evidence of sarcoid (involvement by biopsy ( pulmonary or extrapulmonary)) . Subjects with concurrent extrapulmonary sarcoidosis particularly skin and eye involvement are encouraged to be enrolled. Patients with neurologic sarcoidosis will be excluded.
5. Have FVC > 40 and < 80% of predicted.
6. Have an ATS dyspnea score of > Grade 1.
7. Have been receiving pre-study treatment that includes at least 10 mg/day of prednisone or equivalent dose of corticosteroids as a single agent, and/or methotrexate, or hydroxychloroquine for at least the 3-month period prior to screening. Subjects must be on a stable dose of these meds for > 4 weeks before starting the study medication.
8. Adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) must be used for the duration of the study and should continue such precautions for 6 12 months after receiving the last study infusion.
9. Are considered eligible based on TB screening.
10. Are capable of reading and understanding subject assessment forms and providing written informed consent.
11. Are willing and able to adhere to the study visit schedule and other protocol-specified procedures.

Exclusion Criteria:

Laboratory Exclusion Criteria

1. Hemoglobin: < 8.5 gm/dL
2. Platelets: < 100,000/mm
3. Serum Creatinine: > 1.4
4. Neutrophils: < 1.5 x mm3
5. IgG: < 5.6 mg/dl and IgM: < .55 mg/dl
6. AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
7. Positive Hepatitis B or C serology (Hep B surface antigen and Hep C antibody)

General Safety Exclusion Criteria

1. Previous Treatment with Rituximab (MabThera® / Rituxan®)
2. Previous administration of a treatment with any other therapeutic agent targeted at depleting B cells within 12 months prior to screening.
3. Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
4. Current treatment with TNF inhibitors, cyclosporine, tacrolimus or leflunomide.
5. Treatment with TNF inhibitors within (8 weeks prior to screening), cyclosporine or tacrolimus ( 4 weeks prior to screening) or leflunomide ( 8 weeks prior to screening, or 25 days after cholestyramine washout).
6. Previous treatment within 6 months with IVIg.
7. Parenteral corticosteroids within 4 weeks prior to screening visit.
8. Receipt of live virus or bacterial vaccinations within the 4 weeks before the first dose of the study agent or are expected to receive any live virus or bacterial vaccinations during the trial or up to 3 months after the last dose of the study agent
9. History of severe allergic or anaphylactic reactions associated with the administration of humanized or murine monoclonal antibodies
10. History of New York Heart Association (NYHA) Class III or IV congestive heart failure(CHF)
11. History of severe right-sided heart failure or cor pulmonale
12. Known active bacterial, viral, fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 2 months of screening or oral antibiotics within 2 weeks prior to screening
13. History of recurrent significant infection or history of recurrent bacterial infections
14. History of opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis and aspergilloma, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening
15. History of known infection with human immunodeficiency virus (HIV)
16. Considered ineligible according to the USA-specific TB screening
17. Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation
18. Current signs and symptoms of systemic lupus erythematosus, or severe, progressive, or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic, or cerebral diseases (with the exception of sarcoidosis).
19. Have normal pulmonary function
20. Have any clinical evidence of intracranial lesions.
21. Have an abnormal neurological examination during baseline assessment
22. Have neurosarcoidosis
23. Have a known history of demyelinating disease such as multiple sclerosis or optic neuritis.
24. Concomitant malignancies or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
25. Have poor tolerability of intravenous infusion or lack of adequate venous access for required blood sampling.
26. History of transplanted organ (with the exception of a corneal transplant > 3 months prior to screening.
27. History of substance abuse or dependency, drug or alcohol within 3 years of screening
28. History of primary or secondary immunodeficiency
29. History of psychiatric disorder that would interfere with normal participation in this protocol
30. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
31. Inability to comply with study and follow-up procedures

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adverse events by week 24 and by week 52 that are considered by the investigator to be reasonably or probably related to Rituximab. | 1 year
Change from baseline in 6-minute walk distance at Week 24 and 52. | 1 year

SECONDARY OUTCOMES:
Change in Borg's CR10 dyspnea score before 6 minute walk at weeks 12, 24, and 52 | 1 year
Change in FVC and percent of predicted FVC at weeks 24 and 52 | 1 year
To assess the effect of rituximab on B cell function as measured by markers of these cells in peripheral blood: CD19, CD27, IgD, and CD38 at baseline and weeks 24 and 52 and BAFF and IL-12p40 at baseline and weeks 12, 24, 36 and 52 | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Sweiss NJ, Lower EE, Mirsaeidi M, Dudek S, Garcia JG, Perkins D, Finn PW, Baughman RP. Rituximab in the treatment of refractory pulmonary sarcoidosis. Eur Respir J. 2014 May;43(5):1525-8. doi: 10.1183/09031936.00224513. Epub 2014 Jan 31. No abstract available. PMID 24488568